CLINICAL TRIAL: NCT05356143
Title: A Single-Dose, Partial-Replicate, Pharmacokinetic, and Comparative Bioavailability Study of Rupatadine 10 mg Tablets and Clarinex® 5 mg Tablets Under Fasting Conditions
Brief Title: A Comparative Study of Rupatadine 10 mg Tablets and Clarinex® 5 mg Tablets Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: J. Uriach and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2020-4903 Version: 1.0
Record Dates: First submitted 2021-11-26; First posted 2022-05-02 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Healthy
MeSH Terms: interventions — rupatadine

STUDY DESIGN:
Intervention Model Description: This is an open-label, single-dose, randomized, three-period, two-treatment, threesequence, crossover, PK, partial replicate, and comparative bioavailability study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Sequence 1 (Other): Subjects will take comparator and active drug at different study periods Treatment sequence AAB
  Interventions: Drug: Rupatadine
- Sequence 2 (Other): Treatment sequence ABA
  Interventions: Drug: Rupatadine
- Sequence 3 (Other): Treatment sequence BAA
  Interventions: Drug: Rupatadine

INTERVENTIONS:
Drug: Rupatadine — Oral single dose 10 mg tablet
  Other Names: Pafinur

SUMMARY:
This is an open-label, single-dose, randomized, three-period, two-treatment, threesequence, crossover, PK, partial replicate, and comparative bioavailability study. This study may be conducted in groups. The same protocol requirements and procedures will be followed for each group.

DETAILED DESCRIPTION:
This study will allow for the determination of the PK and intra-subject variability of rupatadine and metabolites. In addition, this study will compare the bioavailability of the rupatadine formulation (Drug Product 1) to a FDA-approved reference product (Clarinex®) (Drug Product 2) as far as the rupatadine metabolite desloratadine, and the derived compounds, is concerned.

Comparative bioavailability between Drug Product 1 and Drug Product 2 will be determined by a statistical comparison of the AUCt, AUCinf, and Cmax parameters for desloratadine (UR-12790), 3-OH desloratadine (UR-12788), 5-OH desloratadine (UR-12767), 6-OH desloratadine (UR-12766), and 3-OH-glucuronide-desloratadine (UR-12335).

ELIGIBILITY:
Inclusion Criteria:

1. Healthy, non-smoking, male and female subjects, 18 years of age or older.
2. BMI ≥19 kg/m2.
3. Females may be of childbearing or non-childbearing potential:

   * Childbearing potential:

     o Physically capable of becoming pregnant
   * Non-childbearing potential:

     * Surgically sterile (i.e., both ovaries removed, uterus removed, or bilateral tubal ligation); and/or
     * Postmenopausal (no menstrual period for at least 12 consecutive months without any other medical cause).
4. QTc ≤450 msec [corrected using Bazett's formula (QTcB)].
5. Willing to use acceptable, effective methods of contraception for the duration of the entire study.
6. Able to tolerate venipuncture.
7. Be informed of the nature of the study and give written consent prior to any study procedure.

Exclusion Criteria:

1. Known history or presence of clinically significant neurologic, hematologic, endocrine, oncologic, pulmonary, immunologic, genitourinary, psychiatric, or cardiovascular disease or any other condition which, in the opinion of the Investigator, would jeopardize the safety of the subject or impact the validity of the study results.
2. Known or suspected carcinoma.
3. Known history or presence of hypersensitivity or idiosyncratic reaction to rupatadine, desloratadine, or any other drug substances with similar activity.
4. Known history or presence of clinically significant angioedema.
5. Known history or presence of clinically significant lactose, galactose, or fructose intolerance.
6. Any acute illness (e.g. cold, acute infection) which is considered significant by the Investigator and that has not resolved within 7 days before the first drug administration.
7. Presence of hepatic or renal dysfunction.
8. Presence of hay fever, seasonal allergy, or rhinitis.
9. Presence of sinusitis.
10. Presence of nasal symptoms (e.g., blocked and/or runny nose).
11. History of atopic allergy (e.g., asthma, urticaria, eczematous dermatitis).
12. History of drug or alcohol addiction requiring treatment.
13. Positive test result for COVID-19 Ag, HIV, Hepatitis B surface Ag, or Hepatitis C Ab.
14. Positive test result for urine drugs of abuse (amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine, methadone, opiates, phencyclidine, and tricyclic antidepressants) or urine cotinine.
15. Difficulty fasting or consuming standard meals.
16. Use of tobacco or nicotine-containing products within 6 months prior to drug administration.
17. Females who:

    * Have used implanted, injected, intravaginal, or intrauterine hormonal contraceptives within 6 months prior to drug administration;
    * Have used oral or transdermal hormonal contraceptives within 21 days prior to drug administration;
    * Are pregnant (serum hCG consistent with pregnancy); or
    * Are lactating.
18. Donation or loss of whole blood (including clinical trials):

    * ≥50 mL and <500 mL within 30 days prior to drug administration;
    * ≥500 mL within 56 days prior to drug administration.
19. Participation in a clinical trial that involved administration of an investigational medicinal product within 30 days prior to drug administration, or recent participation in a clinical investigation that, in the opinion of the Investigator, would jeopardize subject safety or the integrity of the study results.
20. On a special diet within 30 days prior to drug administration (e.g., liquid, protein, raw food diet).
21. Have had a tattoo or body piercing within 30 days prior to drug administration.
22. Have clinically significant findings in vital signs measurements.
23. Have clinically significant findings in a 12-lead ECG.
24. Have clinically significant abnormal laboratory values.
25. Have significant diseases.
26. Have clinically significant findings from a physical examination.
27. Use of any of the following within 30 days prior to drug administration:

    * Antihistamines;
    * CYP3A4 substrates with a narrow therapeutic index (e.g., ciclosporin, tacrolimus, sirolimus, everolimus, cisapride);
    * Drugs known to alter gastrointestinal pH/movement (e.g., cimetidine, omeprazole, ranitidine);
    * Drugs known to prolong QTc;
    * Enzyme-modifying drugs known to induce/inhibit hepatic drug metabolism, specifically CYP 2C9, 2C19, 2D6, and 3A4 (e.g., ketoconazole, itraconazole, fluconazole, posaconazole, voriconazole, clarithromycin, azithromycin, erythromycin, diltiazem, HIV protease inhibitors, nefazodone);
    * Fluoxetine; or
    * Statins.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2021-12-02 (Actual); Primary Completion 2022-01-13 (Actual); Study Completion 2023-01-05 (Actual)

PRIMARY OUTCOMES:
Comparation of drug products | 3 weeks
  To compare the levels of desloratadine (UR-12790) and its related metabolites (UR-2788, UR-12767, UR-12766, UR-12335) after single-dose administration of Drug Product 1 and Drug Product 2 in healthy subjects under fasting conditions

SECONDARY OUTCOMES:
Bioavailability of drug product 1 | 1 week
  To verify the levels of the pre-desloratadine metabolites (UR-12680, UR-12338, UR- 2605, UR-12333, UR-12783) after the administration of Drug Product 1.
Intra-subject variability | 1 week
  To determine the levels of rupatadine (UR-12592) and the intra-subject variability of rupatadine (UR-12592) and its' metabolites after the administration of Drug Product 1.
Number of adverse events | 1 week
  By checking the adverse events ocurring during the study

CONTACTS AND LOCATIONS:
Locations (1):
- Pharma Medica Research Inc., Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Medexus Pharmaceuticals Inc. RupallTM, Rupatadine (as rupatidine fumarate), Tablet 10 mg, Oral Solution 1 mg/mL. Canada: Health Canada; Revised June 2, 2020. — https://www.accessdata.fda.gov/scripts/cder/daf/index.cfm?event=overview.process&ApplNo=021165
- See also: Merck Sharp & Dohme Corp. Highlights of Prescribing Information. Clarinex® (desloratadine) Tablets, RediTabs, and Oral Solution for oral use. USA: FDA; Revised 3/2019. — https://www.accessdata.fda.gov/scripts/cder/daf/